CLINICAL TRIAL: NCT06664983
Title: A Randomized Phase III Clinical Study Comparing the Combination of TPC Regimen With Cadonilimab Against the TPC Regimen Alone in Anti-PD-1 Resistant Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: TPC Combined With Cadonilimab VS. TPC Alone in Anti-PD-1 Resistant Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, XIANG YANQUN, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-581-02
Record Dates: First submitted 2024-10-17; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPC chemotherapy (Active Comparator): NAB-paclitaxel; cisplatin or lobaplatin and capecitabine
  Interventions: Drug: TPC chemotherapy
- Cadonilimab with TPC chemotherapy (Experimental): cadonilimab plus TPC chemotherapy (NAB-paclitaxel, cisplatin or lobaplatin ; and capecitabine
  Interventions: Drug: cadonilimab combined TPC chemotherapy

INTERVENTIONS:
Drug: TPC chemotherapy — The TPC regimen included NAB-paclitaxel administered at a dose of 200 mg/m2 on day 1, cisplatin at a dose of 60 mg/m2 on day 1, and capecitabine at a dose of 1000 mg/m2, taken orally twice a day on days 1 to 14, for each cycle
  Other Names: NAB-paclitaxel, cisplatin, and capecitabine
  Arms: TPC chemotherapy
Drug: cadonilimab combined TPC chemotherapy — Cadonilimab was intravenously given at dose of 10 mg/kg on day 1. The TPC regimen included NAB-paclitaxel administered at a dose of 200 mg/m2 on day 1, cisplatin at a dose of 60 mg/m2 on day 1, and capecitabine at a dose of 1000 mg/m2, taken orally twice a day on days 1 to 14, for each cycle
  Other Names: cadonilimab combined NAB-paclitaxel, cisplatin, and capecitabine
  Arms: Cadonilimab with TPC chemotherapy

SUMMARY:
With the advancement of large-scale phase III clinical studies such as RATIONALE-309, JUPITER-02, and CAPTAIN-1, the GP regimen combined with immunotherapy has become the recommended first-line treatment for recurrent metastatic nasopharyngeal carcinoma. However, patients receiving first-line chemotherapy plus immunotherapy have a median progression-free survival time of only 9.6 to 21.4 months, indicating that disease progression is still inevitable after first-line chemo-immunotherapy in patients with recurrent/metastatic nasopharyngeal carcinoma. Therefore, second or subsequent line treatment options are crucial for the management of patients with recurrent/metastatic nasopharyngeal carcinoma.

In 2021, the International Society for Cancer Immunotherapy reported a multicenter, open-label, single-arm phase II clinical study of cadonilimab in patients with metastatic nasopharyngeal carcinoma who had failed second-line or subsequent chemotherapy. The data showed that among the 20 evaluable patients enrolled, the objective response rate for cadonilimab monotherapy reached 30%, with a disease control rate of 70%, and the median progression-free survival time was 3.71 months. These study results suggest that cadonilimab demonstrates encouraging anti-tumor activity and good safety in patients with metastatic nasopharyngeal carcinoma who have failed second-line or subsequent chemotherapy.

DETAILED DESCRIPTION:
Cadonilimab (AK104) is humanized bispecific antibody that targets to PD-1 and CTLA-4 . Its tetravalent and no Fc binding design contribute to its high binding activity in the tumor microenvironment and improved safety profile . Recent studies have shown encouraging efficacy and manageable toxicity of cadonilimab in several different cancer types. Cadonilimab monotherapy has shown an ORR of 30% and disease control rate (DCR) of 70%, with the median disease-free survival time of 3.71 months in patients with RM-NPC at the second line setting. There is no study available to explore the role of cadonilimab in anti-PD-1 resistant RM NPC patients.

Our previous study prospectively proven the superiority of TPC regimen (paclitaxel, cisplatin, and capecitabine) versus cisplatin and fluorouracil (PF) as induction treatment for patients with stage IVA NPC in NPC patients. Besides, after achieved disease control from TPC regimen induce therapy, capecitabine maintenance therapy significantly improved PFS for patients with newly diagnosed metastatic NPC with tolerate toxic . These results suggest the promising application prospect of TPC regimen in RM-NPC patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.Histopathological diagnosis confirmed as non-keratinizing nasopharyngeal carcinoma.

  2.Confirmed diagnosis of metastatic or recurrent nasopharyngeal carcinoma, not suitable for radical local treatment.

  3.Patients who have failed first-line or subsequent anti-PD-1 antibody immunotherapy (either monotherapy or combination therapy).

  4.Age between 18 and 70 years. 5.Generally good condition, ECOG score of 0-1, with a life expectancy of ≥3 months.

  6.At least one measurable lesion (according to RECIST 1.1); lesions that have been previously irradiated can be considered target lesions if imaging diagnosis clearly shows progression and they are measurable.

  7.Adequate organ and bone marrow function, specifically hemoglobin (HGB) ≥ 80 g/L, white blood cells (WBC) ≥ 4×10^9/L, and platelets (PLT) ≥ 75×10^9/L. Liver function: total bilirubin (TBIL) < 1.5 times the upper limit of normal (ULN), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) < 2.5 times the ULN; serum albumin (ALB) ≥ 28 g/L; if the patient has liver metastases, ALT or AST < 5×ULN; if the patient has liver or bone metastases, alkaline phosphatase (AKP) < 5×ULN. Prothrombin time (PT) international normalized ratio/PTT < 1.5 times the ULN; cardiac function requirement is left ventricular ejection fraction (LVEF) ≥ 50%.

  7.Voluntarily participate and sign the informed consent form, and accept and comply with the study protocol, laboratory tests, follow-ups, etc.

  8.Female subjects of childbearing potential and male subjects with fertile partners must agree to use effective contraception (such as condoms, regularly prescribed contraceptive pills, etc.) from screening until 6 months after the last treatment.

Exclusion Criteria:

* 1.History of hypersensitivity to monoclonal antibodies. 2.Time interval of less than 6 months from the last first-line TPC chemotherapy.

  3.Known history of interstitial pneumonia. 4.Severe infection occurring within 4 weeks prior to the first administration, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia.

  5.Patients who have used aspirin (>325 mg/day) or dipyridamole, ticlopidine, clopidogrel, and cilostazol within 3 weeks prior to medication, or anticoagulants requiring INR monitoring (such as warfarin), or those who have received any blood components and cell growth factor support therapy within 1 week prior to medication.

  6.Active infections requiring systemic treatment. 7.Active hepatitis B (HBV-DNA ≥ 1000 IU/ml) that persists despite treatment, excluding those with cured hepatitis C; significant clinical bleeding symptoms or a clear bleeding tendency within 1 month prior to medication.

  8.Received the last radiotherapy or antitumor treatment within 3 weeks prior to the first administration.

  9.Known history of active tuberculosis or autoimmune diseases. 10.Patients with HIV infection. 11.Presence of other uncontrolled malignancies. 12.Abnormal function of major organs such as the heart, brain, or lungs, or clinical significance of hydronephrosis, ascites, pericardial effusion, or those undergoing thrombolytic therapy.

  13.Pregnant or breastfeeding women. 14.Individuals with personality or mental disorders, or those lacking full civil capacity or having limited civil capacity.

  15.Currently participating in an interventional clinical study treatment, or having received treatment with other investigational drugs within 4 weeks prior to the first administration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-10-21 (Estimated); Study Completion 2026-10-21 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | from the enrollment to disease progression or death from any cause, assessed up to 12 months
  The primary endpoint was PFS, which was assessed as the time from randomization to disease progression per RECIST v1.1 assessed by IRC or death, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No